CLINICAL TRIAL: NCT00006466
Title: Phase I/II Study to Assess the Safety and Efficacy of Low Doses of Beta LT in Patients With Myeloma
Brief Title: Beta Alethine in Treating Patients With Myeloma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: LifeTime Pharmaceuticals (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068280; LIFETIME-LTP-99-01; LIFETIME-IRB-0300203
Record Dates: First submitted 2000-11-06; First posted 2003-10-08 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2002-09

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm; Precancerous Condition
Keywords: monoclonal gammopathy of undetermined significance; isolated plasmacytoma of bone; extramedullary plasmacytoma; refractory multiple myeloma; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell; Precancerous Conditions; Monoclonal Gammopathy of Undetermined Significance | interventions — alethine

INTERVENTIONS:
Drug: beta alethine

SUMMARY:
RATIONALE: Biological therapies such as beta alethine use different ways to stimulate the immune system and stop cancer cells from growing.

PURPOSE: Phase I/II trial to study the effectiveness of beta alethine in treating patients who have myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the antitumor effects of low-dose beta alethine in patients with myeloma or progressive monoclonal gammopathy of undetermined significance.
* Determine the effects of this regimen on anemia, performance status, pain, and delayed-type hypersensitivity (immune response) in these patients.
* Determine the safety of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive beta alethine subcutaneously every 2 weeks for 6 doses. At day 85, patients may receive an additional 12-week course of therapy in the absence of disease progression or unacceptable toxicity. Patients with an apparent complete response receive additional courses.

Patients are followed for 2 weeks.

PROJECTED ACCRUAL: A total of 13-37 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven myeloma

  * Multiple myeloma
  * Indolent myeloma with slowly progressive bone pathology
  * Smoldering myeloma with no bone pathology but a progressive increase in M-protein
  * Solitary myeloma OR
* Diagnosis of evolving monoclonal gammopathy of undetermined significance with increasing M-protein or decreasing hemoglobin level
* Measurable M-protein or Bence Jones protein
* Indolent disease not requiring therapy allowed
* No clinical signs or evidence of active brain involvement or leptomeningeal disease

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 50-100%

Life expectancy:

* At least 4 months

Hematopoietic:

* See Disease Characteristics
* Neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10 g/dL

Hepatic:

* Bilirubin less than 2.0 mg/dL
* Transaminases no greater than 2.5 times upper limit of normal

Renal:

* Creatinine no greater than 2.0 mg/dL
* Creatinine clearance at least 60 mL/min

Cardiovascular:

* No acute changes on electrocardiogram
* No uncontrolled angina, heart failure, or arrhythmia

Other:

* Adequate nutritional status (total protein at least 60.0 g/L, albumin at least 35 g/L)
* HIV negative
* No AIDS
* No active bacterial infection (e.g., abscess) or with fistula
* No history of alcoholism, drug addiction, or psychotic disorders that would preclude study
* No other nonmalignant disease that would preclude study
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior immunotherapy or cytokines

Chemotherapy:

* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas, mitomycin, or high-dose carboplatin)

Endocrine therapy:

* No concurrent corticosteroids

Radiotherapy:

* No prior radiotherapy to greater than 25% of bone marrow

Surgery:

* Recovered from any prior surgery
* No prior solid organ transplantation

Other:

* No other concurrent investigational agent
* No concurrent immunosuppressive agents
* No concurrent anti-inflammatory agents, including aspirin or over-the-counter or prescription nonsteroidal anti-inflammatory drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-08

CONTACTS AND LOCATIONS:
Overall Officials: Suzin Mayerson, PhD, Study Chair — LifeTime Pharmaceuticals
Locations (3):
- United States (3):
  - Emory Clinic, Atlanta, Georgia
  - Victory Over Cancer, Rockville, Maryland
  - St. Vincents Comprehensive Cancer Center, New York, New York